CLINICAL TRIAL: NCT01228851
Title: A Pilot Study of the Effects of Balance Training Using the Wii Balance Board on Balance and Ambulation in Adults With Parkinson's Disease
Brief Title: Balance Training in Parkinson's Disease Using the Wii Balance Board
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Santiago Toledo MD, Rehabilitation Institute of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30775
Record Dates: First submitted 2010-08-31; First posted 2010-10-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Rehabilitation; Balance; Exercise; Parkinson's disease with balance deficits; H&Y 2.5-3
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balance Training (Experimental): Balance training using Wii Fit Balance Board
  Interventions: Other: Balance Training

INTERVENTIONS:
Other: Balance Training — Group balance training sessions three times a week for 8 weeks
  Other Names: Wii (Registered Trademark) Balance Board

SUMMARY:
The purpose of this study is to assess the facilitation of balance in Parkinson's disease (PD) patients using the Nintendo Wii fit, with the ultimate goal of developing a program for function and fitness in this patient population. In this study, PD patients will participate in group exercise classes using the Wii Fit and the effects on balance, postural sway, and quality of life assessed.

DETAILED DESCRIPTION:
The study is a cohort study using outpatients with Parkinson's Disease in Hoen and Yahr Stage 2.5 - 3. Participants will have pre- and post-exercise testing, as well as participate in an 8-week balance-training program.

Subjects Subjects will be recruited from the outpatient clinics (physician, therapy) at the Rehabilitation Institute of Chicago (RIC) as well as the Northwestern Movement Disorders Clinic, through the Department of Neurology. Approximately 20 subjects will be screened for inclusion from these institutions and 12 subjects will be enrolled in the study. (see Power analysis below).

Recruitment Procedures

Potential subjects will be approached by their treating outpatient physician (Physiatrist or Neurologist) or Physical or Occupational Therapist to see if they would be interested in participating in the study. The principal investigator will also send introductory letters to his outpatients at RIC informing them of the study. Letters will only be sent to the PI's patients (Dr. Marciniak, Dr. Toledo). Potential subjects will be educated regarding study procedures, risks and benefits, and privacy risks. Informed consent will be obtained only during initial screening and signed if the patient is interested in proceeding. Eligibility criteria will be screened for (See below). Subjects who lack decisional capacity will not included in the study.

Study Procedures This study will involve an initial visit (Visit 1) for screening and baseline data collection. The therapy/intervention sessions will be held 3 times per week for 8 weeks, (Visits 2 - 25), and there will be 1 post-intervention visit for data collection (Visit 26). Subjects will be reimbursed 11 dollars for parking expenses that will be mailed to them weekly in the form of a check. All visits will take place at Abbott Hall, 3rd floor exercise room and all visits will take approximately 1 ½ hrs.

Visit 1

Following consent, the following baseline measures will be performed:

1. Physician screening with a medical history (including falls in the month prior to the visit) and physical examination
2. Mini Mental Status Examination (MMSE)
3. Hoehn and Yahr Staging
4. Questionnaires:

   1. Activities-Specific Balance Scale
   2. Parkinson's Disease Quality of Life measure (PDQ-8 c. Geriatric Depression Scale.
5. Berg Balance Scale, performed by a trained physical therapist
6. Dynamic Gait Index, performed by the physical therapist
7. Gait and mobility subscales of the UPDRS
8. Sharpened Romberg with eyes open and closed
9. Balance will also be measured using the Wii balance board. Subjects will stand on the board and a gait belt will be placed around their waist. Subjects will have an accelerometer (done via smart phone) clipped to their waist to measure sway, they will stand on the Wii board, and the subject's ability to performing a reaching task will be assessed, as measured by postural sway.

The investigator will remain immediately next to the subject during the testing procedures for safety purposes with the gait belt in place, and a balance bar will also be next to the patient during the testing procedures.

Visits 2- 25 (3x/ week for 8 weeks) (Within 2 weeks of initial testing) The subjects will be seen at the Wirtz Sports Center exercise room. They will participate in 3 Wii balance board games: a marble game, a skiing game, and a bubble game. Each subject will stand on a balance board and participate in each of the 3 games for 10 minutes per game with 10 minutes rest in between each of the games, a total of 30 minutes of balance training time per session. Subjects will have a gait belt in place during the exercises, and will be supervised by a physical therapist or research assistant. Either the Physical therapist or Research Assistant will always be immediately next to the subjects during the training program. A balance bar will also be next to the subject if needed for balance.

Weekly, subjects will be asked about any changes in medications or falls that they may have experienced at home or in the community.

Visit 26

Subjects will seen for follow up assessments within 2 weeks of the final training session and the following tests repeated:

1. Interval history (including falls), exam, Hoehn and Yahr Staging
2. Questionnaires:

   1. Activities-Specific Balance Scale
   2. PDQ-8
   3. Geriatric Depression Scale.
3. Berg Balance Scale
4. Dynamic Gait Index
5. United Parkinson Disease Rating Scale, subscales
6. Sharpened Romberg
7. Wii Balance Board Testing

ELIGIBILITY:
Inclusion Criteria:

1. Adult, 18 years or greater
2. The patient is able to provide informed consent.
3. Definitive Idiopathic Parkinson's Disease as diagnosed by a Neurologist
4. Hoehn and Yahr Stage 2.5-3
5. Able to ambulate at least 150 ft without an assistive device per patient report
6. On stable doses of Parkinson's medications for at least 2 weeks prior to study onset
7. Endurance sufficient to stand at least 20 minutes unassisted per patient report

Exclusion Criteria:

1. Mini Mental Status Exam (MMSE) < 24
2. Anticipated change in Parkinson's medications in the duration of study
3. Uncontrolled orthostasis
4. Symptomatic coronary artery disease
5. Fracture of lower limb within 6 months prior to study onset
6. Other neurologic diagnosis, including Multiple Sclerosis
7. Other vestibular disease
8. Untreated severe depression (depression of greater than or equal 20 on the Geriatric Depression Scale)
9. Acute illness
10. History of, or current, alcohol abuse
11. Significant visual impairment that would inhibit ability to participate in study, with distance vision >20/40
12. Drug induced or inherited Parkinson's Disease
13. Physical therapy within the month prior to study entry
14. Use of the Wii balance board at home as an exercise program
15. Significant camptocormia
16. Physical Therapy during the study duration
17. Any medical condition which the physician investigator determines would compromise the safety of exercise program for the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 8 weeks

SECONDARY OUTCOMES:
Dynamic Gait Index | 8 weeks
Parkinson's Disease QOL Questionnaire (PDQ-8) | 8 weeks
Postural Sway | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States